CLINICAL TRIAL: NCT04569344
Title: COVID-19 and Venous Thromboembolism Risk
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Permanente (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NOACs-1510-32651_enhancement
Record Dates: First submitted 2020-09-25; First posted 2020-09-29 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Venous Thromboembolism; Covid19
MeSH Terms: conditions — Venous Thromboembolism; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Covid-19: Patients with laboratory test positive for SARS-CoV-2 virus
  Interventions: Other: Laboratory test positive for SARS-CoV-2 virus

INTERVENTIONS:
Other: Laboratory test positive for SARS-CoV-2 virus — Exposure/intervention: diagnosis of Covid-19, defined as positive laboratory test for SARS-CoV-2

SUMMARY:
Coronavirus disease 2019 (Covid-19) is now a leading cause of death among U.S. adults. In addition to profound respiratory and multi-organ failure, hypercoagulable states and venous thromboembolism (VTE) have been increasingly reported in patients with severe Covid-19. The aim of this study is evaluate the risk of VTE related to Covid-19 infection in a real-world community-based population.

DETAILED DESCRIPTION:
This is an observational study of adult (age ≥18 years) members enrolled in the Kaiser Permanente Northern California (KPNC) or Kaiser Permanente Southern California (KPSC) integrated healthcare delivery systems during the time period January 1, 2020 through January 31, 2021, (representing the first year of the Covid-19 pandemic) and diagnosed with incident Covid-19. The outcomes will be incident VTE and all-cause death, assessed through February 28, 2021. The primary analysis will describe the rate of post-Covid-19 VTE after index diagnosis. A second analysis will compare the risk of VTE in hospitalized patients with Covid-19 compared with matched hospitalized controls without Covid-19.

ELIGIBILITY:
Inclusion

* Covid-19 diagnosis (defined as date of a positive laboratory test for SARS-CoV-2 virus) during the time period January 1, 2020 to January 31, 2021
* Age >=18 years
* Continuous pharmacy benefits and health plan membership for at least 12 months before the index date

Exclusion

• incomplete information on age and sex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source populations for the study will be adults diagnosed with acute Covid-19 who were enrolled in Kaiser Permanente Northern California or Kaiser Permanente Southern California, two large, integrated healthcare delivery systems in California.
Sampling Method: Non-Probability Sample
Enrollment: 398530 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Acute venous thromboembolism (VTE) | From the date of first positive test for SARS-CoV-2 virus occuring after January 1, 2020, until death, disenrollment from the health system, or the end of the planned outcome assessment (February 28, 2021)
  VTE will be defined as a clinical encounter with evidence of acute VTE, identified by diagnosis codes, +/- radiology procedure codes
Death | From the date of first positive test for SARS-CoV-2 virus occuring after January 1, 2020, until disenrollment from the health system, or the end of the planned outcome assessment (February 28, 2021)
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Margaret C Fang, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Kaiser Permanente Northern California, Oakland, California
  - Kaiser Permanente Southern California, Pasadena, California

IPD SHARING:
Plan to Share IPD: No